CLINICAL TRIAL: NCT06371417
Title: Phase 1b Open-label Basket Trial of RAY121 to Inhibit Classical Complement Pathway in Immunological Diseases (RAINBOW Trial)
Brief Title: Phase 1b Trial of RAY121 in Immunological Diseases (RAINBOW Trial)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAY902CT
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Antiphospholipid Syndrome (APS); Bullous Pemphigoid (BP); Behçet's Syndrome (BS); Dermatomyositis (DM); Immune-mediated Necrotizing Myopathy (IMNM); Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Antiphospholipid Syndrome; Pemphigoid, Bullous; Behcet Syndrome; Dermatomyositis; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAY121 (Experimental): All enrolled patients will receive RAY121 multiple dose
  Interventions: Drug: RAY121

INTERVENTIONS:
Drug: RAY121 — Injection

SUMMARY:
This Phase 1b basket trial will investigate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity and preliminary efficacy of RAY121, a inhibitor of classical complement pathway, after multiple dose administration in patients with immunological diseases such as antiphospholipid syndrome (APS), bullous pemphigoid (BP), Behçet's Syndrome (BS), dermatomyositis (DM), immune-mediated necrotizing myopathy (IMNM) and immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age >= 18 and <=75 at the time of signing informed consent form (except for BP; Age >=18 and <= 85 with Karnofsky score >= 60% at screening)
3. Ability to comply with the study protocol
4. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods
5. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
6. APS cohort: Established primary APS defined by the following criteria (at least one of the laboratory criteria and one of the clinical criteria must be met):

   * Laboratory criteria (aPL profile)

     * Persistently positive lupus anticoagulant (LA) test
     * Persistently positive anticardiolipin (aCL) immunoglobulin G (IgG) isotype
     * Persistently positive anti-beta-2 glycoprotein-1 (aβ2GPI) IgG isotype
   * Clinical criteria

     * Livedoid vasculopathy and presence of skin ulcer
     * Acute/chronic aPL nephropathy
7. BP cohort:

   * 1) Age >= 18 and <= 85 with Karnofsky score >= 60 %
   * 2) Predominant cutaneous lesions
   * 3) Diagnosis with BP with following assessments positive:
   * a Positive direct immunofluorescence, and either
   * b Positive indirect immunofluorescence, or
   * c Positive serology on ELISA for BP180 autoantibody
   * 4) Bullous Pemphigoid Disease Area Index (BPDAI) score >= 20
   * 5) Weekly average of daily Peak Pruritus Numerical Rating Score (PP-NRS) >=4
   * 6) Accept to take photograph of bullous lesions
8. BS cohort:

   * 1) Diagnosed with BS
   * 2) Oral ulcers that occurred at least 3 times in the previous 12 month period
   * 3) Have at least 2 oral ulcers over the 4 weeks prior to screening
   * 4) Have at least 2 oral ulcers at Week 0
   * 5) Have prior treatment with at least 1 non-biologic BS therapy
   * 6) Patients who need systemic therapy as whose oral or mucocutaneous ulcers cannot be adequately controlled by topical therapy
9. DM cohort:

   * 1) Diagnosed with definite or probable inflammatory myopathies and categorized as DM
   * 2) Patients with inadequate response to corticosteroids and/or immune-suppressants or intolerance to DM therapies
   * 3) Manual Muscle Test-8 (MMT-8) score < 142, with at least one abnormality in the following Core Set Measures:

     * Patient Global Activity Visual Analogue Scale (PtGA-VAS) >= 2 cm
     * Physician Global Activity Visual Analogue Scale (PhGA-VAS) >= 2 cm
     * Global extra-muscular activity >= 2 cm
     * At least one muscle enzyme > 1.5 times upper limit of normal (ULN)
     * Health Assessment Questionnaire (HAQ) >= 0.25
   * 4) Moderate to severe DM defined as CDASI activity score > 14
10. IMNM cohort:

    * 1) Clinically Diagnosed with IMNM as anti-HMGCR myopathy or anti-SRP myopathy
    * 2) Creatine kinase (CK) > 1,000 U/L
    * 3) Patients who have an inadequate response to corticosteroids and/or immunosuppressants or intolerance to IMNM therapies
    * 4) MMT-8 score < 142
11. ITP cohort:

    * 1) Confirmed diagnosis of persistent/chronic ITP based on the following criteria:

      * ITP defined per the current guidelines
      * Platelet count <= 30 × 10^9/L on 2 consecutive occasions
    * 2) Lack of an sustained adequate platelet count response to a thrombopoietin receptor agonist and at least one other ITP treatment or a second thrombopoietin receptor agonist (TPO-RA)
    * 3) A history of response with an platelet counts increase more than 20 × 10^9/L from baseline by at least one prior line of therapy

Exclusion Criteria:

1. History of anaphylaxis or hypersensitivity to a biologic agent
2. Active infection requiring systemic antiviral, antibiotics or antifungal
3. Planned surgery during the study
4. Pregnant or breastfeeding, or intending to become pregnant
5. Any serious medical condition or abnormality in clinical laboratory tests that precludes the patient's safe participation in and completion of the study
6. Clinically significant ECG abnormalities
7. Illicit drug or alcohol abuse
8. Clinical diagnosis of autoimmune diseases other than the target disease (except for Sjögren's syndrome in DM and IMNM)
9. Positive for hepatitis B surface antigen
10. Positive for hepatitis C virus antibody
11. Positive for human immunodeficiency virus antibody
12. Evidence of current infection with tuberculosis
13. History of cancer within 5 years
14. Treatment with investigational therapy within 28 days or 5 half-lives
15. Previous and current treatment with anti-C1s antibody at any time
16. Other complement inhibitors within 3 months
17. Patients who receive any treatments which fall into the Prohibited Therapy Criteria
18. Patients with an elevated alanine aminotransferase or aspartate aminotransferase > 1.5 × ULN in combination with an elevated total bilirubin > 1.5 × ULN
19. APS cohort:

    * 1) APS associated with other systemic autoimmune disease
    * 2) Acute thrombosis (arterial or venous acute thrombosis diagnosis) within 30 days before screening
    * 3) Patients with thrombotic APS without any anticoagulation treatment
    * 4) Treatment with prohibited medications
20. BP cohort:

    * 1) Initiation of treatment with or increase in the dose of systemic or topical corticosteroid within 2 weeks
    * 2) Current treatment with a drug that may cause or exacerbate BP unless the dose has been stable
    * 3) Initiation of treatment with topical calcineurin inhibitor, or topical phosphodiesterase (PDE) 4 inhibitor within 7 days
    * 4) Treatment with prohibited medications
21. BS cohort:

    * 1) BS-related active major organ involvement-ocular lesions requiring immunosuppressive therapy, pulmonary (e.g., pulmonary artery aneurysm), vascular (e.g., thrombophlebitis), gastrointestinal (e.g., ulcers along the gastrointestinal tract), and central nervous systems (e.g., meningoencephalitis) manifestations
    * 2) History of venous or arterial thrombosis within 1 year
    * 3) Treatment with prohibited medications
22. DM cohort:

    * 1) PhGA-VAS improvement >= 3, or clinically relevant improvement between screening and baseline
    * 2) Overlap myositis (except for overlap with Sjögren's syndrome), connective tissue disease associated DM, inclusion body myositis, polymyositis, IMNM, juvenile DM or drug-induced myopathy
    * 3) Cancer-associated myositis
    * 4) Significant muscle damage
    * 5) Past history of severe Interstitial lung disease flare, severe non-infectious lung inflammation which required active intervention, or multiple episodes of lung disease
    * 6) Severe respiratory muscle weakness
    * 7) Severe bulbar palsy
    * 8) Treatment with prohibited medications
23. IMNM cohort:

    * 1) PhGA-VAS improvement >= 3, or clinically relevant improvement between screening and baseline
    * 2) Overlap myositis (except for overlap with Sjögren's syndrome), connective tissue disease associated DM, inclusion body myositis, polymyositis, juvenile DM or druginduced myopathy
    * 3) Cancer-associated myositis
    * 4) Significant muscle damage
    * 5) Past history of severe Interstitial lung disease (ILD) flare, severe non-infectious lung inflammation which required active intervention, or multiple episodes of lung disease
    * 6) Severe respiratory muscle weakness
    * 7) Severe bulbar palsy
    * 8) Treatment with prohibited medications
24. ITP cohort:

    * 1) Secondary ITP
    * 2) Clinical diagnosis or history of Myelodysplastic Syndrome or autoimmune hemolytic anemia
    * 3) History of venous or arterial thrombosis within 12 months
    * 4) Patients who experienced major bleeding within 4 weeks
    * 5) Treatment with prohibited medications
    * 6) Any laboratory test results meet either of the following criteria at screening:

      * Hemoglobin <10 g/dL
      * Thyroid-stimulating hormone >= 10 μIU/mL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline to Week 32
  Incidence, severity, and causal relationship of AEs

SECONDARY OUTCOMES:
RAY121 concentration | Baseline to Week 32
  Serum RAY121 concentration
AUCτ | Baseline to Week 32
  Area under the concentration-time curve over a dosing interval (AUCτ)
Cmax | Baseline to Week 32
  Maximum observed serum concentration (Cmax)
Cmin | Baseline to Week 32
  Minimum observed serum concentration (Cmin)
Active C1s | Baseline to Week 32
  Active C1s
Total C1s | Baseline to Week 32
  Total C1s
Complement activity (classical pathway) | Baseline to Week 32
  Complement activity (classical pathway)
Anti-RAY121 antibodies | Baseline to Week 32
  Titer of anti-RAY121 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co.Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (67):
- United States (9):
  - University of California-Irvine, Orange, California
  - Johns Hopkins University, Baltimore, Maryland
  - Northwell Health, LLC PRIME, Lake Success, New York
  - Hospital for Special Surgery, New York, New York
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Amarillo Center for Clinical Research, Amarillo, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Campbelltown Public Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
- AKH - Medizinische Universitaet Wien, Abteilung fuer Klinische Pharmakologie, Vienna, Austria
- Bulgaria (3):
  - Diagnostic Consultation Center CONVEX EOOD, Sofia, Sofia City Province
  - "SHATHD" EAD Sofia, Sofia, Sofia City Province
  - UMHAT "Prof. Dr. St. Kirkovich", AD, Stara Zagora, Stara Zagora Province
- Canada (5):
  - University of Alberta Hospital - Department of Anesthesiology and Pain Medicine, Edmonton, Alberta
  - University of Alberta Hospital - Dermatology, Edmonton, Alberta
  - The Royal Institution for the Advancement of Learning/McGill University, Montreal, Quebec
  - Centre de Rhumatologie de l'Est du Quebec, Rimouski, Quebec
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Croatia (3):
  - Clinical Hospital Center "Sestre Milosrdnice", Zagreb, City of Zagreb
  - University hospital centre Zagreb, Zagreb, City of Zagreb
  - Specialty Hospital Medico, Rijeka, Primorje-Gorski Kotar County
- Sanatorium Profesora Arenbergera, Prague, Prague, Czechia
- France (2):
  - Hopital Lapeyronie,Service d'Immuno Rhumatologie, Montpellier, Occitanie
  - AP-HP Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Klinik und Poliklinik f. Dermatologie, Sachsen, Bundesländer
  - Universitaetsmedizin Goettingen, Göttingen, Göttingen District
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Klinik f Dermatologie, Allergologie u Venerologie, Lübeck, Schleswig-Holstein
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád-Csanád County
  - Semmelweis Egyetem, Budapest
- Italy (3):
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio Dei Tumori "Dino Amadori" - IRST, Meldola, Forlì-Cesena Province
  - Istituto Clinico Humanitas, Milan, Milan Province
  - Ospedale San Giovanni Bosco, Torino, Turin Province
- Japan (8):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Okayama University Hospital, Okayama
- Netherlands (2):
  - University Medical Centre Groningen UMCG, Groningen, Groningen Province
  - UMC Utrecht, Utrecht, Utrecht Province
- Norway (2):
  - Sorlandet sykehus Kristiansand, Kristiansand, Agder County
  - Stavanger Universitetssjukehus, Stavanger, Rogaland County
- Institute Reumatologii I'm. Eleonory Reicher, Warsaw, Masovian Voivodeship, Poland
- Portugal (2):
  - Centro Clinico Academico Braga, Braga, Braga District
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia, Porto District
- Romania (2):
  - Centrul Medical Monza SRL, Bucharest, Bucharest Municipality
  - Oncology Institute Prof. Dr. Ion Chiricuta I.O.C.N., Cluj-Napoca, Cluj
- Spain (7):
  - Clinica Universidad de Navarra, Pamplona, Community of Madrid & Navarre
  - Hospital Universitario Ramon y Cajal, Servicio de Reumatologia, Madrid, Madrid
  - Hospital Universitario 12 de October, Madrid, Madrid
  - Hospital Universitari Vall d'Hebron, Internal Medicine Dept., Barcelona, Province of Barcelona and Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Province Of Córdoba
  - Hospital Universitario Virgen del Rocio, Seville, Province Of Seville
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taichung Veterans General Hospital, Taipei
- Turkey (Türkiye) (2):
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).